CLINICAL TRIAL: NCT02538224
Title: Randomized, Double Blind, Placebo Controlled Clinical Trial of Compare With Doxycycline Plus Ketoprofen Gel in Chronic Periodontitis
Brief Title: Efficacy of Subgingivally Delivered Doxycycline Plus Ketoprofen Gel as an Adjunct to Non-surgical Periodontal Treatment
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Islamic Azad University, Sanandaj (Other)
Responsible Party: Principal Investigator, Amirhossein Farahmand, azadtehran, Islamic Azad University, Sanandaj
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: azadtehran
Record Dates: First submitted 2015-08-20; First posted 2015-09-02 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-06

CONDITIONS: Chronic Periodontitis
Keywords: Periodontitis; doxycycline/ketoprofen topical gel therapeutic
MeSH Terms: conditions — Chronic Periodontitis; Periodontitis | interventions — Doxycycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- experimental(case): group A (Active Comparator): Group A: 2.5%ketoprofen gel + 3 % doxycycline gel which(0.05cc,mixed gel) be put into the periodontal pocket using an insulin syringe;For every 15 days within 3 months .
  Interventions: Drug: 2.5%ketoprofen gel + 3 % doxycycline; Drug: :2.5%ketoprofen gel
- control: group B (Sham Comparator): Group B: 2.5%ketoprofen gel which (0.05cc,gel)be put into the periodontal pocket using an insulin syringe;For every 15 days within 3 months .
  Interventions: Drug: :2.5%ketoprofen gel

INTERVENTIONS:
Drug: 2.5%ketoprofen gel + 3 % doxycycline — GroupA:(0.05cc, mixed gel) be put into the periodontal pocket using an insulin syringe.
  Intervention category Treatment: drugs
  Other Names: Experimental
  Arms: experimental(case): group A
Drug: :2.5%ketoprofen gel — GroupB:2.5%ketoprofen gel which be inserted into the periodontal pocket using an insulin syringe .
  Other Names: control

SUMMARY:
Objectives: The aim of the present clinical study was to evaluate the efficacy of doxycyline 3% plus ketoprofen 2.5% as an adjunct to scaling and root planing in the treatment of chronic periodontitis(early-modearte). Material and Methods: 20 systemically healthy, chronic periodontitis patients were included in the study.The Patients were selected on the basis of having chronic periodontitis with periodontal pocket depths of more than 4mm on at least two teeth in mandibular molar area; Periodontal parameters (plaque, bleeding on probing and pocket depth) were recorded at baseline and every 15 days for 3 months. Oral hygiene instructions were given that included brushing twice- daily, (Using the Bass brushing technique for at least 2 minutes ), Randomly divided two groups,Test group: was treated by scaling and root planing Followed by local delivery of doxycycline 3%+ ketoprofen 2.5%, While the control group: was treated by scaling and root planing along with ketoprofen 2.5%; and was administered to the both groups every 15 days for 3 months, repeated. Every 15 days once periodontal parameters were assessed, and at the end of 3 months, evaluated the clinical parameters changes.

DETAILED DESCRIPTION:
Source of Data In this 8 month follow up, longitudinal intervention study, a total of 20patients (9 males and 11 females, Age range: 30-50 years) with chronic periodontitis were selected from the outpatient section of the Department of Periodontics, Islamic Azad University Dental School of Tehran /Iran. The study met the criteria of the Helsinki Declaration of1975, revised in 2008. The survey plan was reviewed and sanctioned, approved by the ethics commission of the Institutional Ethical Committee and Review Board of the Deputy of Research, School of Dentistry. All subjects received oral and written explanation of the intent of the survey and signed an informed consent after receiving detailed information about the purpose, the benefits, and the possible risks associated with the trial. The study was conducted from October 2012 to November 2013. The study was registered at the Iranian registry of clinical trials (IRCT), registration code: IRCT2014050717587N2.

Selection Criteria Patients meeting all of the following criteria were included in the study: aged between 30 and 45 years; 20 natural teeth present; clinical and radiographic signs of moderate (clinical attachment level of 2 to 3mm); probing depth (PD) of >4 mm; no periodontal treatment the previous 6 months; and willingness to comply with the study protocol.

Patients were excluded from the study if they met one or more of the following criteria: 1) existing systemic disease that may influence the severity or progression of periodontitis; taking medications that may influence the periodontium (e.g., non-steroidal anti-inflammatory drugs) or other medicines (antibiotic) within the 6 months preceding the beginning of the study; concurrent or planned orthodontic treatments; planned extensive dental restorations; patients with cavitated caries; pregnancy or lactation; mouth rinses during the entire period of the study; hypersensitive to doxycycline or ketoprofen; smoking.

Grouping Criteria Patients received scaling and root planing on first visit in accordance with the one stage full-mouth debridement protocol + polishing; the therapeutic endpoint was defined as a clean root surface void of visible or clinically detectable remnants of biofilm or calculus. After 2 weeks (debridement), was applied into all periodontal pockets with PD of ≥4 mm using a syringe with a blunt canula. The canula was inserted to the base of the periodontal pocket and gel was applied 0/5 ml on each side of the mandible. After patient enrollment by an examiner; using blocked randomization with a block size of 4 and an allocation ratio of 1:1 Block randomization was chosen to prevent too much variability in the number of patients randomized and ensure a reasonably steady flow of patients to each treatment group, Allocation cover was ensured by using container and labeling that did not reveal the content of the trial drug packages who was blind to the therapist and the clinical examination. Patients were randomly assigned to either the A or B group, while mandibular arches are each divided into two parts (left and right sections) with 100 sites in both groups.

In the A group, was treated by scaling and root planing (SRP) followed by local delivery of doxycycline 3%+ ketoprofen 2.5%, while the B group was treated by scaling and root planing along with ketoprofen 2.5%; and was administered to the both groups every 15 days for 3 months. After treatment, patients were given thorough oral hygiene instructions, the trial gel for local application contained ketoprofen gel (2.5% Sanofi Pharmaceutical plant construction in France) + 3 % doxycycline (Kharazmi Pharmaceutical manufacture in Iran) in the group (A), another group (B) ketoprofen 2.5%gel was used. After treatment, patients were given thorough oral hygiene instructions and were asked to use dentifrice sodium fluorides (Crest cavity protection) and to finish from using any mouthwashes during the course of the study. The subjects were given careful instructions in self-performed plaque-control measures: twice-daily tooth brushing using the Bass brushing technique with a soft toothbrush and a regular fluoride containing toothpaste and once-daily Interdental cleaning using dental floss. Clinical parameters, including Plaque Index (PI) (18), sulcus bleeding index (19). Probing depth (PD) and clinical attachment level (CAL) were recorded at baseline (before the SRP) and at 0, 15,30,45,60 days and 3 months. William's periodontal probe was used to standardize the measurement of clinical parameters. All pre- and post-treatment clinical parameters were recorded by an examiner who was masked to the type of treatment received by the patients while another clinician provided treatment for both groups. All pre- and post-treatment clinical parameters were recorded by an examiner who was masked to the type of treatment received by the patients while another clinician provided treatment for both groups.

ELIGIBILITY:
Inclusion Criteria:

* adult patients,
* older than 18 years old,
* systemically healthy, and
* having at least 20 teeth.

Exclusion Criteria:

* patients with cavitated caries,
* no periodontal pockets larger than 4 mm,
* orthodontic appliances or removable prostheses,
* allergies to cetylpyridinium or CHX,
* use of antibiotics and anti-inflammatory drugs in the past 3 months that might alter normal gingival health,
* oral prophylaxis outside of study;
* use of oral chlorhexidine products or participation in an oral rinse study within 3 months prior to baseline examination,
* pregnancy or lactation,
* smoking.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-07; Primary Completion 2014-02 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Reduction of pocket depth | 15 days

SECONDARY OUTCOMES:
Reduction of bleeding on probing | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: amirhossein farahmand, assoc prof, Principal Investigator — azad tehran

IPD SHARING:
Plan to Share IPD: No